CLINICAL TRIAL: NCT00194935
Title: A Phase II Trial of Weekly Topotecan As Consolidation Therapy in Ovarian Cancer Patients After Initial Chemotherapy
Brief Title: Weekly Topotecan Therapy in Patients With Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-636
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Cancer of the Ovary
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan

INTERVENTIONS:
Drug: Topotecan

SUMMARY:
The purpose of this study is to find out the safety and feasibility of weekly topotecan consolidation therapy in patients with ovarian cancer.

DETAILED DESCRIPTION:
Patients with Stage IIIC and IV optimally-debulked ovarian cancer will be treated with 6 cycles (every 3 weeks) of carboplatin (AUC 5) and paclitaxel (175 mg/m2). Patients who demonstrate a complete clinical response to this regimen will then be treated with topotecan consolidation (4 mg/m2 weekly x 8 weeks for one cycle followed by a break in the 9th week) for a maximum of 3 cycles. Primary endpoints will be toxicity and the determination of the appropriate dose, schedule, and duration of topotecan for further consolidation trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histopathologic diagnosis of epithelial ovarian cancer.
* Patients must have completed front-line chemotherapy and be clinically NED (CA 125 <35, negative CT scan, negative physical exam).
* Patients may have a second look laparoscopy, however, there must be no gross disease present (microscopic disease or pathologically negative).
* Patients must not have had other myelosuppressive therapy within four weeks of initiating topotecan therapy.
* Topotecan treatment must begin within 10 weeks following last cycle of initial chemotherapy.
* Patients may have had only one prior chemotherapy regimen.

Exclusion Criteria:

* Patients with a concomitant malignancy other than squamous cell or basal cell skin cancer.
* Patients who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2003-02; Study Completion 2006-08

PRIMARY OUTCOMES:
The objective of this study is to evaluate the safety and feasibility of weekly topotecan consolidation therapy in patients with epithelial ovarian cancer.

SECONDARY OUTCOMES:
To determine the efficacy (Progression free survival) of weekly topotecan as consolidation therapy in ovarian cancer patients who are clinically NED or have microscopic disease only after first-line chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caputo, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medcial College of Cornell University, New York, New York, United States